CLINICAL TRIAL: NCT02406495
Title: Clinical Performance of Habitual Wearers of Bioclear 1-day Lenses When Refitted With Biomedics 1-day Extra for 1 Week
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EX-MKTG-58
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Results first posted 2016-05-03 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Myopia; Hyperopia
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- filcon IV 1 and ocufilcon D (Experimental): Habitual wearers of filcon IV 1 sphere lenses refitted with asphere ocufilcon D lenses.
  Interventions: Device: filcon IV 1; Device: ocufilcon D

INTERVENTIONS:
Device: filcon IV 1 — contact lens
Device: ocufilcon D — contact lens

SUMMARY:
Open label, 1-week daily disposable, dispensing study

DETAILED DESCRIPTION:
Evaluate the clinical performance of habitual wearers of FILCON IV 1 sphere lenses when refitted with ocufilcon D asphere for 1 week of daily disposable wear.

ELIGIBILITY:
Inclusion Criteria:

* Is between 18 and 40 years of age (inclusive)
* Has had a self-reported visual exam in the last two years
* Is an adapted Avaira sphere contact lens wearer (at least 1 week in Avaira sphere)
* Has a contact lens spherical prescription between + 2.25 to - 8.00 (inclusive)
* Has a spectacle cylinder up to 0.75D in each eye.
* Can achieve best corrected spectacle distance visual acuity of 20/25 (0.10 logMAR) or better in each eye.
* Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses.
* Has clear corneas and no active ocular disease
* Has read, understood and signed the information consent letter.
* Patient contact lens refraction should fit within the available parameters of the study lenses.
* Is willing to comply with the wear schedule (at least 5 days per week, > 8 hours/day assuming there are no contraindications for doing so).
* Is willing to comply with the visit schedule

Exclusion Criteria:

* Is not a habitual wearer of Avaira sphere lenses
* Has a CL prescription outside the range of the available parameters of the study lenses.
* Has a spectacle cylinder ≥1.00D of cylinder in either eye.
* Has a history of not achieving comfortable CL wear (5 days per week; > 8 hours/day)
* Has contact lens best corrected distance vision worse than 20/25 (0.10 logMAR) in either eye.
* Presence of clinically significant (grade 2-4) anterior segment abnormalities
* Presence of ocular or systemic disease or need of medications which might interfere with contact lens wear.
* Slit lamp findings that would contraindicate contact lens wear such as:

  * Pathological dry eye or associated findings
  * Pterygium, pinguecula, or corneal scars within the visual axis
  * Neovascularization > 0.75 mm in from of the limbus
  * Giant papillary conjunctivitis (GCP) worse than grade 1
  * Anterior uveitis or iritis (past or present)
  * Seborrheic eczema, Seborrheic conjunctivitis
  * History of corneal ulcers or fungal infections
  * Poor personal hygiene
* Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
* Has aphakia, keratoconus or a highly irregular cornea.
* Has Presbyopia or has dependence on spectacles for near work over the contact lenses.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Montés-Mico, OD MPhil PhD, Principal Investigator — Optometry Research Group (GIO) Optics Department, University of Valencia
Locations (1):
- Optometry Research Group (GIO) Optics Department, University of Valencia, Valencia, Spain

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Participants: Habitual wearers of (FILCON IV 1) sphere lenses refitted with asphere ocufilcon D lenses.
  filcon IV 1: contact lens
  ocufilcon D: contact lens
Period: Overall Study
Arm/Group | Overall Participants
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Participants
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.92 (5.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 9

OUTCOME MEASURES:

1. Secondary Outcome: Visual Acuity - Filcon IV 1 and Ocufilcon D
Description: Visual acuity for filcon IV 1 assessed at baseline and ocufilcon D assessed at 1 week using logMAR chart (a logMAR of 0.0=20/20 in Snellen notation and negative values indicate better visual acuity).
Time Frame: Baseline and 1 Week
Measure: Mean (Standard Deviation); unit: LogMAR
Groups:
- Filcon IV 1; Ocufilcon D: Habitual wearers of (FILCON IV 1) sphere lenses refitted with asphere ocufilcon D lenses.
  filcon IV 1: contact lens
  ocufilcon D: contact lens
Arm/Group | Filcon IV 1 | Ocufilcon D
Number analyzed (Participants) | 40 | 40
LogMAR
  OD | 0 (0) | 0 (0)
  OS | 0 (0) | 0 (0)
  Binocular | -0.01 (0.03) | -0.01 (0.04)

2. Secondary Outcome: Comfort (Subjective Ratings) - Filcon IV 1 and Ocufilcon D
Description: Subjective ratings for comfort for filcon IV 1 assessed at baseline and ocufilcon D assessed at 1 week. (Scale 0-10, 0=could feel, 10=cannot feel).
Time Frame: Baseline and 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Filcon IV 1 | Ocufilcon D
Number analyzed (Participants) | 40 | 40
units on a scale
  Comfort on insertion | 7.4 (1.1) | 8.1 (1.3)
  Comfort prior to removal | 7.3 (1.4) | 8.1 (1.3)
  Comfort overall | 7.3 (1.3) | 8.1 (1.4)

3. Primary Outcome: Lens Fit, Centration - Filcon IV 1 and Ocufilcon D
Description: Lens fit, centration for filcon IV 1 assessed at baseline and ocufilcon D assessed at 1 week. Scale: optimum, decentration acceptable, and decentration unacceptable
Time Frame: Baseline and 1 Week
Measure: Number; unit: percentage of eyes
Groups:
- Filcon IV 1 OD (Oculus Dexter); Filcon IV 1 OS (Oculus Sinister); Ocufilcon D OD (Oculus Dexter); Ocufilcon D OS (Oculus Sinister): Habitual wearers of (FILCON IV 1) sphere lenses refitted with asphere ocufilcon D lenses.
  filcon IV 1: contact lens
  ocufilcon D: contact lens
Arm/Group | Filcon IV 1 OD (Oculus Dexter) | Filcon IV 1 OS (Oculus Sinister) | Ocufilcon D OD (Oculus Dexter) | Ocufilcon D OS (Oculus Sinister)
Number analyzed (Participants) | 40 | 40 | 40 | 40
percentage of eyes
  Optimum | 58 | 70 | 98 | 98
  Decentration acceptable | 43 | 30 | 3 | 3
  Decentration unacceptable | 0 | 0 | 0 | 0

4. Primary Outcome: Lens Fit, Post-blink Movement - Filcon IV 1 and Ocufilcon D
Description: Lens fit, post-blink movement for filcon IV 1 assessed at baseline and ocufilcon D assessed at 1 week.
  (Scale 0-4, 0=Insufficient, unacceptable movement, 1=Minimal, but acceptable movement, 2=Optimal movement, 3=Moderate, but acceptable movement, 4=Excessive, unacceptable movement).
Time Frame: Baseline and 1 Week
Measure: Number; unit: percentage of eyes
Groups:
- Filcon IV 1 OD; Filcon IV 1 OS; Ocufilcon D OD; Ocufilcon D OS: Habitual wearers of (FILCON IV 1) sphere lenses refitted with asphere ocufilcon D lenses.
  filcon IV 1: contact lens
  ocufilcon D: contact lens
Arm/Group | Filcon IV 1 OD | Filcon IV 1 OS | Ocufilcon D OD | Ocufilcon D OS
Number analyzed (Participants) | 40 | 40 | 40 | 40
percentage of eyes
  0=Insufficient, unacceptable movement | 0 | 0 | 0 | 0
  1=Minimal, but acceptable movement | 10 | 10 | 0 | 0
  2=Optimal movement | 23 | 18 | 10 | 10
  3=Moderate, but acceptable movement | 65 | 70 | 90 | 90
  4=Excessive, unacceptable movement | 3 | 3 | 0 | 0

5. Primary Outcome: Lens Fit, Lens Tightness - Filcon IV 1 and Ocufilcon D
Description: Lens fit, lens tightness for filcon IV 1 assessed at baseline and ocufilcon D assessed at 1 week.
  Scale 0%-100% continuous scale 0% - Falls from cornea without lid support 50% - Optimum 100% - No movement
Time Frame: Baseline and 1 Week
Measure: Mean (Standard Deviation); unit: percentage of mean lens tightness
Arm/Group | Filcon IV 1 | Ocufilcon D
Number analyzed (Participants) | 40 | 40
percentage of mean lens tightness
  OD | 49.1 (5.9) | 50.1 (0.79)
  OS | 48.9 (5.2) | 50.0 (1.9)

6. Primary Outcome: Lens Fit, Overall Fit Acceptance - Filcon IV 1 and Ocufilcon D
Description: Lens fit, overall fit acceptance for filcon IV 1 assessed at baseline and ocufilcon D assessed at 1 week. Scale 0-4, 0=Should not be worn, 4=Perfect.
Time Frame: Baseline and 1 Week
Measure: Number; unit: percentage of eyes
Arm/Group | Filcon IV 1 OD | Filcon IV 1 OS | Ocufilcon D OD | Ocufilcon D OS
Number analyzed (Participants) | 40 | 40 | 40 | 40
percentage of eyes
  Should not be worn | 0 | 0 | 0 | 0
  Borderline but acceptable | 0 | 0 | 0 | 0
  Min. acceptable | 0 | 0 | 0 | 0
  Not perfect but OK | 38 | 35 | 0 | 0
  Perfect | 63 | 65 | 100 | 100

7. Secondary Outcome: Dryness (Subjective Ratings) - Filcon IV 1 and Ocufilcon D
Description: Subjective ratings of dryness for filcon IV 1 assessed at baseline and ocufilcon D assessed at 1 week. (Scale 0-10, 0=dryness, 10=no dryness).
Time Frame: Baseline and 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Filcon IV 1 | Ocufilcon D
Number analyzed (Participants) | 40 | 40
units on a scale
  Dryness during day | 7.2 (1.3) | 8.0 (1.5)
  Dryness prior to removal | 7.3 (1.3) | 8.0 (1.5)
  Overall dryness | 7.3 (1.3) | 8.1 (1.5)

8. Secondary Outcome: Handling (Subjective Ratings) - Filcon IV 1 and Ocufilcon D
Description: Subjective ratings of handling for filcon IV 1 assessed at baseline and ocufilcon D assessed at 1 week. (Scale 0-10, 0=very difficult to handle, 10=very easy to handle).
Time Frame: Baseline and 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Filcon IV 1 | Ocufilcon D
Number analyzed (Participants) | 40 | 40
units on a scale | 7.4 (1.2) | 8.2 (1.3)

9. Secondary Outcome: Vision Satisfaction (Subjective Ratings) - Filcon IV 1 and Ocufilcon D
Description: Subjective ratings of vision satisfaction for filcon IV 1 assessed at baseline and ocufilcon D assessed at 1 week. (Scale 0-10, 0=dissatisfied, 10=very satisfied).
Time Frame: Baseline and 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Filcon IV 1 | Ocufilcon D
Number analyzed (Participants) | 40 | 40
units on a scale | 7.5 (1.3) | 8.2 (1.3)

10. Secondary Outcome: Lens Preference (Subjective Ratings) - Filcon IV 1 and Ocufilcon D
Description: Subjective ratings of participant's lens preference for either filcon IV 1 or ocufilcon D on comfort, dryness, handling, vision, and overall. Forced choice: filcon IV 1 or ocufilcon D.
Time Frame: 1 Week
Measure: Number; unit: percentage of participants
Arm/Group | Filcon IV 1 | Ocufilcon D
Number analyzed (Participants) | 40 | 40
percentage of participants
  Comfort | 20 | 80
  Dryness | 20 | 80
  Handling | 20 | 80
  Vision | 20 | 80
  Overall | 20 | 80

11. Secondary Outcome: Lens Satisfaction, Comfort - Filcon IV 1 and Ocufilcon D
Description: Lens satisfaction of comfort for filcon IV 1 assessed at baseline and ocufilcon D assessed at 1 week. Scale 1-4, 1=completely satisfied, 4=completely dissatisfied.
Time Frame: Baseline and 1 Week
Measure: Number; unit: percentage of participants
Arm/Group | Filcon IV 1 | Ocufilcon D
Number analyzed (Participants) | 40 | 40
percentage of participants
  Completely Satisfied | 20 | 60
  Somewhat Satisfied | 68 | 35
  Somewhat Dissatisfied | 13 | 5
  Completely Dissatisfied | 0 | 0

12. Secondary Outcome: Lens Satisfaction, Dryness - Filcon IV 1 and Ocufilcon D
Description: Lens satisfaction of dryness for filcon IV 1 assessed at baseline and ocufilcon D assessed at 1 week. Scale 1-4, 1=completely satisfied, 4=completely dissatisfied.
Time Frame: Baseline and 1 Week
Measure: Number; unit: percentage of participants
Arm/Group | Filcon IV 1 | Ocufilcon D
Number analyzed (Participants) | 40 | 40
percentage of participants
  Completely Satisfied | 20 | 60
  Somewhat Satisfied | 65 | 35
  Somewhat Dissatisfied | 15 | 5
  Completely Dissatisfied | 0 | 0

13. Secondary Outcome: Lens Satisfaction, Handling - Filcon IV 1 and Ocufilcon D
Description: Lens satisfaction of handling forfilcon IV 1 assessed at baseline and ocufilcon D assessed at 1 week. Scale 1-4, 1=completely satisfied, 4=completely dissatisfied.
Time Frame: Baseline and 1 Week
Measure: Number; unit: percentage of participants
Arm/Group | Filcon IV 1 | Ocufilcon D
Number analyzed (Participants) | 40 | 40
percentage of participants
  Completely Satisfied | 23 | 60
  Somewhat Satisfied | 65 | 38
  Somewhat Dissatisfied | 13 | 3
  Completely Dissatisfied | 0 | 0

14. Secondary Outcome: Lens Satisfaction, Vision - Filcon IV 1 and Ocufilcon D
Description: Lens satisfaction of vision for filcon IV 1 assessed at baseline and ocufilcon D assessed at 1 week. Scale 1-4, 1=completely satisfied, 4=completely dissatisfied.
Time Frame: Baseline and 1 Week
Measure: Number; unit: percentage of participants
Arm/Group | Filcon IV 1 | Ocufilcon D
Number analyzed (Participants) | 40 | 40
percentage of participants
  Completely Satisfied | 23 | 60
  Somewhat Satisfied | 65 | 38
  Somewhat Dissatisfied | 13 | 3
  Completely Dissatisfied | 0 | 0

15. Secondary Outcome: Lens Satisfaction, Overall - Filcon IV 1 and Ocufilcon D
Description: Lens satisfaction overall for filcon IV 1 assessed at baseline and ocufilcon D assessed at 1 week. Scale 1-4, 1=completely satisfied, 4=completely dissatisfied.
Time Frame: Baseline and 1 Week
Measure: Number; unit: percentage of participants
Arm/Group | Filcon IV 1 | Ocufilcon D
Number analyzed (Participants) | 40 | 40
percentage of participants
  Completely Satisfied | 20 | 60
  Somewhat Satisfied | 68 | 35
  Somewhat Dissatisfied | 13 | 5
  Completely Dissatisfied | 0 | 0

ADVERSE EVENTS:
Time Frame: From dispense up to one week for each study lenses
Arm/Group | Overall Participants
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study.

There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

The investigators will not be permitted to publish or present at scientific meetings results obtained from the clinical study without prior written consent from the sponsor.